CLINICAL TRIAL: NCT02591927
Title: Reappraisal of Glucose-insulin-potassium Therapy in Acute St-segment Elevation Myocardial Infarction by Pre-hospital Administration
Brief Title: Reappraisal of GIK in Acute STEMI by Pre-hospital Administration
Acronym: REAGIK-STEMI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Pier Giorgio Masci, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 32003B_159727
Record Dates: First submitted 2015-10-28; First posted 2015-10-30 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; glucose-insulin-potassium
MeSH Terms: conditions — Myocardial Infarction | interventions — glucose-insulin-potassium cardioplegic solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucose-Insulin-Potassium (Active Comparator): Rackley's Glucose-Insulin-Potassium formula consisting of 30% glucose (300 mg/L), 50 units of regular insulin per liter and 80 mEqu of KCL per liter.
  Interventions: Drug: Glucose-Insulin-Potassium
- Glucose 5% (Placebo Comparator): Glucose 5%
  Interventions: Drug: Glucose 5%

INTERVENTIONS:
Drug: Glucose-Insulin-Potassium — Rackley's GIK formula by continuous I.V. infusion at 1.5 ml/Kg/hour for 12 hours (about 100 ml/hour for a 70 kg patient).
  Other Names: GIK
  Arms: Glucose-Insulin-Potassium
Drug: Glucose 5% — Glucose 5% (Placebo) by continuous I.V. infusion at 1.5ml/kg/hour for 12 hours (about 100 ml/hour for 70 Kg patient)
  Other Names: Placebo
  Arms: Glucose 5%

SUMMARY:
The purpose of this study is:

1. to assess whether pre-hospital glucose-insulin-potassium (GIK) administration in acute STEMI patients would reduce infarct size and ischemia/reperfusion damage using comprehensive tissue characterization by cardiovascular magnetic resonance (CMR) at an early post-infarction phase.
2. to explore the putative cardioprotective mechanisms of pre-hospital GIK administration

DETAILED DESCRIPTION:
Background - After an acute ST-segment elevation myocardial infarction (STEMI), early and successful myocardial reperfusion with primary percutaneous coronary intervention (PCI) is the most effective strategy for reducing the infarct size and improving clinical outcome. The process of restoring blood flow to the ischemic myocardium, however, can induce injury per se, paradoxically increasing the extent of final infarction (i.e., reperfusion injury). Research has been focusing for years on a strategy to effectively counteract reperfusion injury and, thereby, reduce the final infarct size with salutary effects on clinical outcome. Robust experimental evidences support Glucose-Insulin-Potassium (GIK) as an effective cardioprotective agent being capable to metabolically protect the myocardium against ischemia and ischemia/reperfusion injury. These benefits are clearly related to the time that GIK is administered in the course of cardiac ischemia, with effectiveness increasing with early administration. However, clinical trials in the reperfusion era have lost the opportunity to translate the beneficial effects seen in the laboratory to the clinical setting, because of the unacceptably prolonged delay from the onset of ischemic symptoms to GIK administration. A properly-designed prospective trial with double-blinded randomization to placebo or GIK in the out-of-hospital setting would straightforwardly overcome this limitation, thereby providing convincing evidences in favor or disfavor of GIK treatment. Notable, GIK is an un-expensive compound, and upon the verification of its efficacy, GIK treatment would be ready for primetime clinical application with matchless cost/effectiveness profile.

Aims

1. to assess whether pre-hospital GIK administration in acute STEMI patients would reduce infarct size and ischemia/reperfusion damage using comprehensive tissue characterization by cardiovascular magnetic resonance (CMR) at an early post-infarction phase.
2. to explore the putative cardioprotective mechanisms of pre-hospital GIK administration

Methods - The investigators will conduct a single-center randomized, placebo-controlled, double-blinded trial for testing the efficacy of pre-hospital GIK administration in patients with acutely reperfused STEMI. The pre-specified primary end-point is the reduction of infarct size, as quantitated by late gadolinium enhancement CMR in the early post-infarction phase. Major secondary end-points are: 1) reduction of ischemia/reperfusion injury quantitated by CMR, and 2) investigation of the putative cardioprotective mechanisms ofGIK treatment in subjects with acute STEMI.

Outlook: The investigators study results, if positive, will persuade the scientific community to reconsider pre-hospital GIK treatment as adjunctive to primary PCI in acute STEMI patients and revitalize the field of metabolism-based cardioprotection. They will illustrate by which mechanisms cardioprotection is achieved in the clinical setting, prompting large prospective multicentre trials to test the efficacy of pre-hospital GIK administration on hard clinical end-points.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with the diagnosis of acute STEMI
2. age≥ 18
3. informed consent for study participation.

Exclusion Criteria evaluated during ambulance transport to primary PCI center:

1. end-stage renal failure requiring dialysis,
2. prior MI or coronary revascularization (PCI or CABG),
3. active malignances,
4. Pregnancy,
5. Hemodynamic instability (systolic blood pressure <100mmHg or significant pulmonary congestion defined as O2 saturation <90% on ambient air at pulso-oxymetry)

Exclusion Criteria evaluated after hospital admission at the primary PCI center (all patients will be re-evaluated for study continuation):

1. total ischemic time more than 8 hours (from symptoms onset to infarct-related artery mechanical re-opening)
2. evidence at diagnostic angiograms of TIMI flow-grade >1 of infarct-related artery or significant epicardial collaterals to the ischemic myocardium at risk (Rentrop flow-grade >1),
3. moderate-to-severe renal failure (estimated glomerular filtration rate < 30 ml/min/1.73 m2 by Cockcroft-Gault formula) and
4. urgent CABG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2016-02; Primary Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Infarct size quantified by Late Gadolinium Enhancement using Cardiovascular Magnetic Resonance | 12 to 72 hours after the acute event

SECONDARY OUTCOMES:
The severity of ischemia/reperfusion injury (myocardial edema, microvascular obstruction and myocardial hemorrhage) | 12 to 72 hours after the acute event
  The of ischemia/reperfusion injury will be assessed by multiparametric CMR
Major Adverse Cardiovascular Events | at 7-day, 30-day, 4-month and at 1-year follow-up
Post-infarction Remodeling | 4-month follow-up
  Adverse post-infarction remodeling is defined as increase of LV end-systolic volume more than 15% between the first CMR (12 to 72 hours after the acute event) and second CMR (4-month after the acute event)

CONTACTS AND LOCATIONS:
Overall Officials: Pier-Giorgio Masci, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois; Juerg Schwitter, MD, Study Director — Centre Hospitalier Universitaire Vaudois; Pierre Vogt, MD, Study Chair — Centre Hospitalier Universitaire Vadois; Eric Eeckhout, MD, Study Chair — Centre Hospitalier Universitaire Vaudois; Juan-Fernando Iglesias, Study Chair — Centre Hospitalier Universitaire Vaudois; Olivier Muller, Study Chair — Centre Hospitalier Universitaire Vaudois; Olivier Hugli, Study Chair — Centre Hospitalier Universitaire Vaudois; Fabrice Dami, Study Chair — Centre Hospitalier Universitaire Vaudois; Pierre Monney, Study Chair — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois - CHUV, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Grossman AN, Opie LH, Beshansky JR, Ingwall JS, Rackley CE, Selker HP. Glucose-insulin-potassium revived: current status in acute coronary syndromes and the energy-depleted heart. Circulation. 2013 Mar 5;127(9):1040-8. doi: 10.1161/CIRCULATIONAHA.112.130625. No abstract available. PMID 23459576
- [Background] Selker HP, Beshansky JR, Sheehan PR, Massaro JM, Griffith JL, D'Agostino RB, Ruthazer R, Atkins JM, Sayah AJ, Levy MK, Richards ME, Aufderheide TP, Braude DA, Pirrallo RG, Doyle DD, Frascone RJ, Kosiak DJ, Leaming JM, Van Gelder CM, Walter GP, Wayne MA, Woolard RH, Opie LH, Rackley CE, Apstein CS, Udelson JE. Out-of-hospital administration of intravenous glucose-insulin-potassium in patients with suspected acute coronary syndromes: the IMMEDIATE randomized controlled trial. JAMA. 2012 May 9;307(18):1925-33. doi: 10.1001/jama.2012.426. Epub 2012 Mar 27. PMID 22452807